CLINICAL TRIAL: NCT03172143
Title: Mesenteric Sparing Versus High Ligation Ileocolic Resection for the Prevention of Recurrent Crohn's Disease
Brief Title: Mesenteric Sparing for the Prevention of Recurrent Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual not met
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amy L Lightner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-008144
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Crohn Disease
Keywords: Ileocolic; Crohn's; Terminal ilium; Ileocecal
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients with Crohns Disease will be randomized in a 1:1 ratio for mesenteric sparing versus high ligation of the ileocolic artery when performing an ileocolic resection for Crohn's disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenteric sparing ileocolic resection (Active Comparator): Ileocolic resection without removal of the lymph nodes in the mesentery.
  Interventions: Procedure: Mesenteric Sparing Ileocolic Resection
- High ligation ileocolic resection (Active Comparator): Ileocolic resection with removal of lymph nodes in the mesentery
  Interventions: Procedure: High Ligation Ileocolic Resection

INTERVENTIONS:
Procedure: Mesenteric Sparing Ileocolic Resection — In this resection, the mesentery will be spared, or left in situ during resection.
  Arms: Mesenteric sparing ileocolic resection
Procedure: High Ligation Ileocolic Resection — In this resection, a "high ligation" is performed, where the feeding vessel is taken at its origin in order to take sufficient mesentery and lymph nodes with the colon specimen.
  Arms: High ligation ileocolic resection

SUMMARY:
The purpose of this study is to determine if taking an increased sampling of mesentery (fatty tissue next to the intestine) and lymph nodes at the time of the subject's ileocolic resection prevents a 4-6 month recurrence of Crohn's disease at the site of the new connection.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory disease of the intestinal tract with an unknown etiology and an unknown cure. The characteristic transmural inflammation can progress to refractory inflammatory disease, stricturing disease, and fistulizing disease - all potential indications for surgery when medical management has been exhausted. An important tenant to remember is that surgery is not curative but is rather an adjunct to maximal medical therapy.

One third of patients with CD will require a major abdominal resection within 5 years of their diagnosis, and two-thirds will ultimately require operative management at least once during the course of their disease. Unfortunately, surgery for CD is not curative and disease recurrence is common with 62% having endoscopic recurrence at six months, and 80% and 30% of patients having endoscopic and clinical recurrence, respectively, at one year. A third of these patients will require a re-operation at 10 years and up to 80% will require an additional operation by 15 years. This undoubtedly leads to an increased probability of malabsorption syndrome and decreased quality of life.

A significant volume of research has been conducted in attempt to determine how to prevent postoperative recurrence of CD following an ileocolic resection. Some studies have focused on the timing of resuming postoperative medical therapy. Others have looked at surgical technique at the time of ileocolic resection including anatomic configuration of the anastomosis and performing a stapled versus handsewn anastomosis.

There is recent evidence to suggest that the mesentery is actively involved in the ongoing disease process. The investigators plan to investigate if taking additional mesentery affects postoperative recurrence to support these findings.

ELIGIBILITY:
Inclusion Criteria:

1. Residents of the United States
2. Isolated ileocolic Crohn's disease without evidence of perforation
3. Concurrent therapies with corticosteroids, 5-aminosalicylic acid (5-ASA) drugs, thiopurines, methotrexate (MTX), antibiotics, and anti-tumor necrosis factor (TNF) therapy are permitted
4. All patients should have undergone a colonoscopy and CT enterography in last 3 months to assess severity of disease
5. Have no contraindications to magnetic resonance (MR) evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Medically refractory disease or inability to tolerate ongoing medical therapy

Exclusion Criteria:

1. Inability to give informed consent.
2. Patients undergoing repeat ileocolic resection
3. Patients with concurrent disease in other locations (e.g., proximal stricturing of the small bowel, fistulizing disease to the sigmoid colon) requiring additional operation intervention beyond an ileocolic resection
4. Clinically significant medical conditions within the six months before administration of Mesenchymal Stem Cells (MSCs): e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient
5. Specific exclusions;

   a. Evidence of hepatitis B, C, or HIV
6. History of cancer including melanoma (with the exception of localized skin cancers)
7. Emergent indication for an operation
8. A resident outside the United States
9. Pregnant or breast feeding.
10. History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
11. Inability to follow up at Mayo Clinic at 3 to 4 and 12 months for postoperative imaging and endoscopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Number of Subjects who have Recurrence of Crohn's Disease at 6 Months | 6 months after surgery
  Subjects who have endoscopic or histologic evidence of recurrence

SECONDARY OUTCOMES:
Differences in gross and histologic margins with each approach following surgery. | 1 year after surgery
  Determine the need for restarting immunosuppressive medication within the first year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Lightner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No